CLINICAL TRIAL: NCT06612970
Title: A Phase 1a, Randomized, Double-blind, Placebo-controlled, Single Dose-escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HB0056 in Adult Healthy Subjects.
Brief Title: A Study to Evaluate Single-dose of HB0056 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: HB0056-HV-01-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: HB0056

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- HB0056 dose group 1 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 2 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 3 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 4 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 5 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 6 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- HB0056 dose group 7 (Active Comparator): HB0056 single dose
  Interventions: Drug: HB0056
- Matching placebo for each dose group (Placebo Comparator): placebo, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HB0056 — HB0056 Injection
  Other Names: Targeting TSLP and IL-11 IgG1-type Bispecific Antibody
  Arms: HB0056 dose group 1; HB0056 dose group 2; HB0056 dose group 3; HB0056 dose group 4; HB0056 dose group 5; HB0056 dose group 6; HB0056 dose group 7
Drug: Placebo — Placebo
  Other Names: No other invention name
  Arms: Matching placebo for each dose group

SUMMARY:
The aim of this study is to investigate the safety and tolerability of HB0056 in healthy subjects following single-dose.

DETAILED DESCRIPTION:
This is a single-dose escalation study of HB0056 to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of HB0056.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects age ≥ 18 and ≤ 55 years.
* Body Mass Index (BMI) ≥ 18 and ≤ 32 kg/m².
* Normal ECG, blood pressure, respiratory rate, temperature, and heart rate, unless the investigator considers any abnormality to be not clinically significant.
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease.
* Current or history of malignancy. • Family history of premature Coronary Heart Disease (CHD)
* History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
* Pregnant or Breasting feeding subject. Women with a positive pregnancy test .
* Further exclusions criteria applied.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with drug related adverse events (AEs) | Up to 2700 hours
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational drug

SECONDARY OUTCOMES:
Cmax | Up to 2700 hours
  The maximum measured concentration of the analysis in plasma.
AUC0-infinity | Up to 2700 hours
  The area under the concentration-time curve of the analysis in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Cory Sellwood, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No